CLINICAL TRIAL: NCT07336082
Title: Somatosensory Training Versus Exercise Therapy in Awake Bruxism: A Randomized Controlled Trial
Brief Title: Somatosensory Training Versus Exercise Therapy in Awake Bruxism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, GulOznur KARABICAK, Assoc Prof, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-15189967-050.04-2500084155
Record Dates: First submitted 2025-12-19; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Bruxism
Keywords: orofacial pain; somatosensory awareness; exercise therapy; awake bruxism; sensorimotor training; neuroplasticity; physical therapy
MeSH Terms: conditions — Bruxism; Facial Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three parallel groups: somatosensory awareness-based training, jaw and posture exercise therapy, or a wait-list control group. Each group is followed concurrently, and outcomes are compared between groups over time.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the interventions, participants and treating physiotherapists cannot be blinded to group allocation. However, all outcome assessments are performed by an independent assessor who is blinded to treatment allocation. Data analysis is also conducted by a researcher who is not involved in treatment delivery and is blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Somatosensory Awareness Training Group (Experimental): Participants assigned to this group will receive a somatosensory retraining and patient education program based on CRAFTA principles. The intervention focuses on tactile and proprioceptive stimulation, body awareness, and body schema-oriented techniques, including tasks such as two-point discrimination training, light touch awareness, mirror-based posture observation, and self-monitoring of parafunctional behaviors. No conventional strengthening or mobility exercises will be provided. Participants will complete daily awareness-based home tasks, and adherence will be monitored weekly through brief structured follow-ups conducted by a research assistant.
  Interventions: Other: Somatosensory Awareness-Based Training
- Jaw and Posture Exercise Group (Active Comparator): Participants in this group will receive a structured physiotherapy program based on previously published protocols. The intervention includes jaw mobility and relaxation exercises, postural alignment and scapular stabilization exercises, and cervical stretching and strengthening exercises. Participants will attend supervised face-to-face sessions twice weekly for four weeks and will also receive a home exercise booklet.
  Interventions: Other: Jaw exercise therapy
- Wait-List Control Group (Other): Participants in the wait-list group will not receive any active intervention during the first four weeks but will continue their usual daily routines. They will be assessed at the same time points as the intervention groups to allow comparison of natural symptom progression. After completion of the primary endpoint assessment, participants in this group will be offered an active intervention according to clinical need.
  Interventions: Other: Wait-List Control

INTERVENTIONS:
Other: Jaw exercise therapy — Participants assigned to this group receive a structured jaw and posture exercise therapy program delivered by a physiotherapist. The intervention consists of supervised face-to-face sessions twice per week over a 4-week period, combined with a home exercise program performed on non-supervised days.
  The program includes jaw mobility and relaxation exercises, postural correction and stabilization exercises, and cervical region exercises. In addition, manual therapy techniques are applied as clinically indicated, including ischemic trigger point therapy, cervical joint mobilization, and intraoral manual techniques. Each treatment session lasts approximately 40-45 minutes. Adherence to the home exercise program is monitored throughout the intervention period.
  Other Names: exercise therapy
  Arms: Jaw and Posture Exercise Group
Other: Somatosensory Awareness-Based Training — Participants in this group receive an individualized somatosensory awareness-based training program designed to target altered sensory perception and body schema related to the face and jaw. The intervention focuses on laterality recognition, body schema representation, and tactile discrimination, including two-point discrimination-based tasks.
  No conventional exercise therapy or manual therapy techniques are provided in this group. The training is delivered using a flexible, patient-specific approach, supported by structured guidance materials aimed at increasing daily awareness and self-monitoring of somatosensory experiences. Participant adherence and engagement are monitored through regular follow-up and self-report tracking.
  Other Names: Somatosensory training; Sensorimotor awareness training
  Arms: Somatosensory Awareness Training Group
Other: Wait-List Control — Participants allocated to the wait-list control group do not receive any active treatment during the initial study period and continue their usual daily activities. All outcome assessments are conducted at the same time points as the intervention groups. After completion of the assessment phase, participants in this group are offered exercise therapy according to clinical need.
  Arms: Wait-List Control Group

SUMMARY:
Awake bruxism (daytime teeth clenching or jaw tension) is a common condition that can cause jaw pain, facial pain, muscle fatigue, and reduced quality of life. Although current treatments often focus on the jaw muscles and posture, recent research suggests that changes in the brain's sensory processing may also play an important role in bruxism-related pain.

This randomized controlled trial aims to compare two physiotherapy-based treatment approaches with a wait-list control group in adults with awake bruxism. Participants will be randomly assigned to one of three groups: (1) somatosensory awareness-based training, (2) jaw and posture exercise therapy, or (3) a wait-list control group.

The somatosensory training program focuses on improving body awareness and sensory perception of the face and jaw, while the exercise program includes jaw mobility, postural alignment, and cervical exercises. Both active interventions will be delivered over a 4-week period. Participants will be assessed at baseline, immediately after treatment, and during follow-up to evaluate changes over time.

The main outcome of this study is orofacial pain intensity. Secondary outcomes include jaw function, sensory processing, muscle structure, oral parafunctional behaviors, and oral health-related quality of life. The results of this study may help improve physiotherapy-based treatment strategies for people with awake bruxism by addressing both physical and sensory aspects of the condition.

DETAILED DESCRIPTION:
Awake bruxism is a repetitive jaw muscle activity occurring during wakefulness and is frequently associated with orofacial pain, muscle fatigue, functional limitations, and reduced oral health-related quality of life. Increasing evidence suggests that bruxism-related pain cannot be fully explained by peripheral mechanisms alone and that central nervous system processes, including maladaptive neuroplasticity and somatosensory cortical reorganization, may play a key role in symptom persistence. Distortions in somatosensory processing, such as impaired tactile acuity, altered laterality recognition, and disrupted facial emotion recognition, have been reported in individuals with chronic orofacial pain.

This single-blind, parallel-group, randomized controlled pilot trial aims to investigate whether a somatosensory awareness-based training program leads to greater improvements in pain, function, and somatosensory processing compared with a conventional jaw and posture exercise program and a wait-list control group in individuals with awake bruxism.

The study will be conducted at the Physiotherapy and Rehabilitation Unit and the Faculty of Dentistry of Aydın Adnan Menderes University. Participant recruitment is planned between December 2025 and September 2026. Eligible participants will be adults aged 18-45 years with a diagnosis of awake bruxism confirmed by an expert dentist using the Standardised Tool for the Assessment of Bruxism (STAB) and DC/TMD Axis I criteria. Additional inclusion criteria include self-reported daytime clenching behavior, baseline orofacial pain intensity of at least 5/10, and the presence of at least one measurable somatosensory impairment identified during clinical or digital assessment. Individuals with severe disability (GCPS Grade IV), systemic inflammatory or neurological disorders, recent jaw-related treatments, or conditions that may interfere with participation will be excluded.

Following baseline assessment (T0), participants will be randomly allocated in a 1:1:1 ratio to one of three groups using stratified block randomization based on age and sex. Allocation concealment will be ensured using sequentially numbered, sealed opaque envelopes managed by an independent research assistant. Due to the nature of the interventions, participant and therapist blinding will not be possible; however, all outcome assessments and data analyses will be performed by assessors blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 45 years
* Clinical diagnosis of awake bruxism confirmed using standardized diagnostic criteria (STAB and DC/TMD Axis I)
* Presence of at least one measurable somatosensory alteration confirmed at baseline using digital and clinical assessments
* Self-reported daytime jaw clenching or parafunctional activity
* Baseline orofacial pain intensity of ≥5/10 on a Visual Analog Scale (VAS)
* Chronic pain graded as GCPS Grades I-III according to DC/TMD Axis II (Turkish validated version)
* Willingness to comply with the study protocol and attend scheduled treatment sessions
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* GCPS Grade IV (high disability level)
* Presence of systemic inflammatory, neurological, or rheumatological disorders
* Diagnosis of severe chronic pain conditions unrelated to bruxism
* Use of occlusal splints or participation in jaw, neck, or facial therapy within the past 3 months
* Psychiatric disorders or cognitive impairment that could interfere with study participation
* Pregnancy, due to potential effects on joint laxity and postural parameters

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Orofacial Pain-Related Disability | Baseline, Week 4 (post-intervention), Week 6, Week 12
  Orofacial pain-related disability will be assessed using the Craniofacial Pain and Disability Inventory (CF-PDI). The CF-PDI is a self-reported questionnaire evaluating pain-related functional limitations, psychosocial impact, and disability. The Craniofacial Pain and Disability Inventory (CF-PDI) total score ranges from 0 to 100, with higher scores indicating greater pain-related disability.
Orofacial Pain Intensity | Baseline, Week 4 (post-intervention), Week 6, Week 12
  Orofacial pain intensity will be assessed using a 0-10 Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Participants will rate their current orofacial pain intensity at the time of assessment.

SECONDARY OUTCOMES:
Mandibular Range of Motion | Baseline, Week 4 (post-intervention), Week 6, Week 12
  Mandibular range of motion will be assessed using standardized clinical measurements, including maximum mouth opening, lateral excursion (right and left, averaged), and protrusion, recorded in millimeters. Higher values indicate greater mandibular mobility.
Masseter Muscle Thickness | Baseline, Week 12
  Masseter muscle thickness will be assessed using ultrasound imaging and recorded in millimeters (mm). Changes in muscle thickness over time will be evaluated as an indicator of structural and neuromuscular adaptation. No a priori assumption will be made regarding the direction of change.
Oral Parafunctional Behaviors | Baseline, Week 4 (post-intervention), Week 12
  The Oral Behaviors Checklist (OBC) assesses the frequency of oral parafunctional behaviors. The total score ranges from 0 to 84, with higher scores indicating more frequent oral behaviors.
Facial Emotion Recognition Accuracy | Baseline, Week 4 (post-intervention), Week 6, Week 12
  Facial emotion recognition will be assessed using a standardized computerized task. The primary metric will be accuracy (%), with higher values indicating better emotion recognition performance.
Oral Health-Related Quality of Life | Baseline, Week 4 (post-intervention), Week 12
  Oral health-related quality of life will be evaluated using the Oral Health Impact Profile-14 (OHIP-14). The Oral Health Impact Profile-14 (OHIP-14) total score ranges from 0 to 56, with higher scores indicating worse oral health-related quality of life.
Bruxism severity | Baseline, Week 4 (post-intervention), Week 12
  Bruxism severity will be assessed using the Bruxism Severity Questionnaire (BSQ), which evaluates the frequency and impact of awake bruxism-related behaviors and symptoms. The Bruxism Status Questionnaire (BSQ) is a 20-item yes/no questionnaire developed to support the clinical evaluation of bruxism. The BSQ is used to provide descriptive background information to assist expert clinicians in confirming the presence of bruxism. Individual item responses will be recorded; no validated total severity score is assumed. The questionnaire will be used for exploratory purposes only.
Mandibular Function | Baseline, Week 4 (post-intervention), Week 6, Week 12
  Mandibular functional mobility will be assessed by measuring maximum mouth opening, lateral excursions, and protrusion using standardized clinical procedures.
Facial Emotion Recognition - Accuracy | Baseline, Week 4 (post-intervention), Week 6, Week 12
  Facial emotion recognition will be assessed using a standardized computerized task.
  The primary outcome will be accuracy (% of correctly identified emotions). Higher values indicate better emotion recognition performance.
Facial Emotion Recognition Response Time | Baseline, Week 4 (post-intervention), Week 6, Week 12
  Facial emotion recognition will be assessed using a standardized computerized task. The primary metric will be response time (seconds) required to correctly identify facial emotions, with lower values indicating faster responses.
Laterality Recognition Accuracy | Baseline, Week 4, Week 6, Week 12
  Laterality recognition will be assessed using a computerized left-right judgment task involving facial and upper extremity images.
  Accuracy (% correct responses) will be recorded. Higher values indicate better laterality recognition.
Laterality Recognition Reaction Time | Baseline, Week 4 (post-intervention), Week 6, Week 12
  Reaction time (seconds) required to make correct left-right judgments will be recorded.
  Lower values indicate faster laterality processing.
Two-Point Discrimination Threshold | Baseline; Week 4; Week 6; Week 12
  Tactile spatial discrimination will be assessed using a standardized two-point discrimination test. The minimum distance (in millimeters) at which two distinct points are perceived as separate will be recorded. Lower values indicate better tactile discrimination.
Light Touch Detection | Baseline; Week 4; Week 6; Week 12
  Light touch sensation will be assessed using standardized clinical testing. The outcome will reflect the participant's ability to detect light tactile stimuli, according to the study protocol. Higher scores indicate better light touch sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Gul Oznur KARABICAK, PhD, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydin Adnan Menderes University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Unit, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly at this stage. The dataset contains detailed clinical and somatosensory assessments, and data sharing is restricted due to ethical approvals and participant consent limitations.
  De-identified data may be made available upon reasonable request after publication, subject to additional ethical approval.

REFERENCES:
- [Background] Soares-Silva L, de Amorim CS, Magno MB, Tavares-Silva C, Maia LC. Effects of different interventions on bruxism: an overview of systematic reviews. Sleep Breath. 2024 Jun;28(3):1465-1476. doi: 10.1007/s11325-023-02961-7. Epub 2024 Jan 4. PMID 38177829
- [Background] Ainoosah S, Farghal AE, Alzemei MS, Saini RS, Gurumurthy V, Quadri SA, Okshah A, Mosaddad SA, Heboyan A. Comparative analysis of different types of occlusal splints for the management of sleep bruxism: a systematic review. BMC Oral Health. 2024 Jan 5;24(1):29. doi: 10.1186/s12903-023-03782-6. PMID 38182999
- [Background] Fernandez-de-Las-Penas C, Von Piekartz H. Clinical Reasoning for the Examination and Physical Therapy Treatment of Temporomandibular Disorders (TMD): A Narrative Literature Review. J Clin Med. 2020 Nov 17;9(11):3686. doi: 10.3390/jcm9113686. PMID 33212937
- [Background] Uchima Koecklin KH, Aliaga-Del Castillo A, Li P. The neural substrates of bruxism: current knowledge and clinical implications. Front Neurol. 2024 Oct 1;15:1451183. doi: 10.3389/fneur.2024.1451183. eCollection 2024. PMID 39410996
- [Background] Kluskens TJ, Kessler PA, Jansma BM, Kaas A, van de Ven V. Neural Correlates of Tooth Clenching in Patients with Bruxism and Temporomandibular Disorder-Related Pain. J Oral Facial Pain Headache. 2023 Spring;37(2):139-148. doi: 10.11607/ofph.3091. PMID 37389840
- [Background] 8. von Piekartz, H., Paris-Aliaga, A., & La Touche, R. (2019). Bruxism and temporomandibular disorders: The role of somatosensory representation distortions in the trigeminal system. Musculoskeletal Science and Practice, 42, 102073. https://doi.org/10.1016/j.msksp.2019.102073
- [Background] 7. Moseley, G. L. (2007). Reconceptualising pain according to modern pain science. Physical Therapy Reviews, 12(3), 169-178. https://doi.org/10.1179/108331907X223010
- [Background] von Piekartz H, Bleiss S, Herzer S, Hall T, Ballenberger N. Does combining oro-facial manual therapy with bruxism neuroscience education affect pain and function in cases of awake bruxism? A pilot study. J Oral Rehabil. 2024 Sep;51(9):1692-1700. doi: 10.1111/joor.13740. Epub 2024 Jun 18. PMID 38894567
- [Background] La Touche R, Cuenca-Martinez F, Suso-Marti L, Garcia-Vicente A, Navarro-Morales B, Paris-Alemany A. Tactile trigeminal region acuity in temporomandibular disorders: A reliability and cross-sectional study. J Oral Rehabil. 2020 Jan;47(1):9-18. doi: 10.1111/joor.12870. Epub 2019 Aug 26. PMID 31394008
- [Background] 4. Osiewicz, M., Lobbezoo, F., Bracci, A., & Manfredini, D. (2024). From bruxism to somatosensory changes and back: A narrative review on the bidirectional link between orofacial pain and cortical reorganization. Frontiers in Oral Health, 5, 1374090. https://doi.org/10.3389/froh.2024.1374090
- [Background] 3. Paris, A. J., Piekartz, H. v., Rinne, P., & Tardif, C. (2021). Altered brain activation in patients with temporomandibular disorders: Evidence from functional imaging studies. Journal of Oral Rehabilitation, 48(6), 685-696. https://doi.org/10.1111/joor.13144
- [Background] Lobbezoo F, Ahlberg J, Glaros AG, Kato T, Koyano K, Lavigne GJ, de Leeuw R, Manfredini D, Svensson P, Winocur E. Bruxism defined and graded: an international consensus. J Oral Rehabil. 2013 Jan;40(1):2-4. doi: 10.1111/joor.12011. Epub 2012 Nov 4. PMID 23121262
- [Background] Manfredini D, Ahlberg J, Aarab G, Bender S, Bracci A, Cistulli PA, Conti PC, De Leeuw R, Durham J, Emodi-Perlman A, Ettlin D, Gallo LM, Haggman-Henrikson B, Hublin C, Kato T, Klasser G, Koutris M, Lavigne GJ, Paesani D, Peroz I, Svensson P, Wetselaar P, Lobbezoo F. Standardised Tool for the Assessment of Bruxism. J Oral Rehabil. 2024 Jan;51(1):29-58. doi: 10.1111/joor.13411. Epub 2023 Feb 10. PMID 36597658